CLINICAL TRIAL: NCT02786238
Title: Cognitive and Self-regulatory Mechanisms Of Obesity Study
Acronym: COSMOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University (Other)
Collaborators: Kent State University (Other); Case Western Reserve University (Other); University of Minnesota (Other); Drexel University (Other); University of Oklahoma (Other); Cherokee Nation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AS-15-46
Record Dates: First submitted 2016-04-12; First posted 2016-05-30 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Behavioral Treatment (SBT) (Active Comparator): For the Standard Behavioral Treatment (SBT) condition, participants will participate in the standard behavioral weight loss programming, which utilizes strategies from existing obesity treatments (e.g., the Diabetes Prevention Program). These features include the following: 1) nutritional education, 2) diet and physical activity, 3) expectations for daily self-monitoring of calorie intake and activity, 4) stimulus control, behavior shaping, behavior analysis, and relapse prevention strategies, and 5) social support.
  Interventions: Behavioral: Standard Behavioral Treatment (SBT)
- Acceptance-Based Treatment (ABT) (Experimental): The Acceptance-Based Treatment (ABT) group will receive most features listed in the SBT arm as well as unique ABT training designed to help individuals increase awareness of their cognitive and affective experiences, and the following exercises: 1) identifying weight-related goals from personal life values (e.g., health) and connecting these values to day-to-day eating, 2) increasing awareness of moment-by-moment behavior choices, 3) tolerating aversive internal states that include eating-related states as well as affective states such as stress, sadness, and anxiety (i.e., "urge-surfing"). These strategies that have been empirically tested and found to be effective in the NIH-funded Mind Your Health RCT (R21DK080430).
  Interventions: Behavioral: Acceptance-Based Treatment (ABT)

INTERVENTIONS:
Behavioral: Standard Behavioral Treatment (SBT) — See description of treatment arm.
  Arms: Standard Behavioral Treatment (SBT)
Behavioral: Acceptance-Based Treatment (ABT) — See description of treatment arm. **Cherokee Nation members receive only the ABT intervention as they are in an open, feasibility trial and are not randomized.**
  Arms: Acceptance-Based Treatment (ABT)

SUMMARY:
This study will be the first clinical trial to examine the impact of two different weight loss interventions on novel mechanisms that promote obesity and impede its successful treatment, including cognitive function and self-regulatory factors. The results will provide important data about how impaired cognitive function and/or self-regulation promote obesity and how different weight loss treatments may differentially impact these factors; this information will be used to identify promising cognitive and self-regulatory treatment targets for preventing further obesity development and for maintaining weight loss.

DETAILED DESCRIPTION:
This K23 award will allow Dr. Misty Hawkins, a clinical psychologist with expertise in behavioral medicine and obesity, to further develop into an independent investigator proficient in physiological, neuropsychological, and self-regulatory research methods and interventions that will allow her to study novel mechanisms of and treatments for obesity maintenance. She has a career interest in intervening on the neuropsychological factors related to obesity. Her research goal is to identify novel cognitive and self-regulatory mechanisms of obesity in this pilot trial which can then be targeted in larger randomized controlled trials (RCTs) to reduce obesity development or to maintain weight loss. Obesity continues to be a global epidemic, yet successful interventions for obesity are rare, with 80% of individuals in treatment programs being unsuccessful at achieving long-term weight loss. The training and research activities in this K23 application will allow her to examine the complexities of physiological dysregulation, cognitive deficits, and self-regulatory failure in an obesity treatment study. The application proposes an intensive, 5-year program of mentored research and formal training activities to enhance Dr. Hawkins' skills and experience in: 1) basic research on and assessment of cognitive function; (2) assessment of obesity-related physiological changes; (3) research with patient populations; (4) advanced assessment of self-regulation (SR); and (5) the conduct of randomized clinical trials and advanced statistics. In the long term, Dr. Hawkins will apply these translational research skills to study targeted cognitive and self-regulation interventions as potentially effective treatments for persons with obesity who may exhibit cognitive deficits or chronic self-regulatory failure. The research component of this career development award is a clinical trial examining the impact of two different weight loss treatments on physiological markers, cognition, self-regulation, and health behaviors in 96 obese persons. The specific aims are to: 1) Confirm that baseline obesity-related physiological dysregulation is linked to cognitive deficits, poorer self-regulation, and obesogenic behaviors, 2) Demonstrate that the two treatment groups have improvements in biomarkers, cognition, SR, and obesogenic behaviors, less weight gain, and greater weight loss, and 3) Evaluate whether the acceptance-based treatment (ABT) group has greater improvements in biomarkers, cognition, SR, and obesogenic behaviors, less weight gain, and greater weight loss than the standard behavioral treatment group (SBT) from pre- to post-treatment and 1-year follow-up. Oklahoma State University and its research partner Oklahoma University Health Sciences Center provide exceptional environments for Dr. Hawkins to gain the skills needed to achieve her goals. The training component uses academic resources including the College of Arts and Sciences and the Department of Psychology. Dr. Hawkins' mentors are highly regarded scientists in the areas of obesity, neuropsychology, psychophysiology, nutrition, and patient-oriented research.

**An open trial arm of ABT was added to the study in September 2016 to test feasibility of ABT among members of Cherokee Nation. This arm is entitled POWER-UP: Pilot Of WEight Reduction in Underserved Populations. Glucose is the only biomarker being measured in POWER-UP.

ELIGIBILITY:
Inclusion Criteria:

* >21 years old
* <65 years old
* BMI > 27
* BMI < 52
* Attended Information/Recruitment session
* **For Cherokee Nation arm of the study only, participants must endorse Native American/American Indian racial identity (POWER-UP).

Exclusion Criteria:

* Age out of stated range
* BMI out of stated range
* Physician says physical activity is contraindicated (won't sign off) or participant meets the criteria on the Physical Activity Readiness Questionnaire (PARQ) for need a physician signature and doesn't obtain one.
* History of bariatric surgery or planning to get surgery over next 12 months
* Pregnant, planning to become pregnant over next 12 months
* Currently breastfeeding
* Failure of Independence (a family member/friend enrolling in study)
* History or current serious eating disorder pathology
* Current severe depression or suicidal ideation
* Current severe anxiety
* History or current substance use disorder
* History of hypomanic or manic episode
* History of psychotic episode
* History of neurological disorder or head injury (e.g., stroke, epilepsy, loss of consciousness >10 min)
* Recent significant weight loss
* Current Type I Diabetes
* Medications or disease that impact weight (e.g., mirtazapine, prednisone, dexamethasone, dronabinol, megestrol, Cushing's syndrome). The exclusion of persons with hypothyroidism was discontinued given very high base rates in recruitment sample. We will run sensitivity analyses by those with and without hypothyroidism.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
% Weight Loss Post-Treatment | 6 months after baseline
  The percentage of weight loss at treatment completion (6 months after baseline).
% Weight Loss at Follow-up | One year after baseline
  The percentage of weight loss at one year after baseline (6 months post-treatment).

SECONDARY OUTCOMES:
Change in Insulin Levels | Baseline to 6-months and Baseline to one-year
  The change in insulin at 6 months and 1 year after baseline.
Change in Fasting Glucose | Baseline to 6-months and Baseline to one-year
  The change in fasting glucose at 6 months and 1 year after baseline.
Change in Hemoglobin A1C | Baseline to 6-months and Baseline to one-year
  The change in fasting Hemoglobin at 6 months and 1 year after baseline.
Change in C-Reactive Protein | Baseline to one-year
  The change in C-Reactive Protein at 1 year after baseline.
Change in Tumor Necrosis Factor-Alpha | Baseline to one-year
  The change in Tumor Necrosis Factor-Alpha at 1 year after baseline.
Change in Interleukin-6 | Baseline to one-year
  The change in Interleukin-6 at 6 months and 1 year after baseline.
Change in Cognitive Function | Baseline to 6-months and Baseline to one-year
  Cognitive function measured using the NIH Toolbox - Cognitive Battery
Change in Self-Regulation | Baseline to 6-months and Baseline to one-year
  Self-regulation measured using two self-report questionnaires and two behavioral tasks. Scores on these tasks will be converted to z-scores and then aggregated into one measure.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hawkins MAW, Colaizzi J, Gunstad J, Hughes JW, Mullins LL, Betts N, Smith CE, Keirns NG, Vohs KD, Moore SM, Forman EM, Lovallo WR. Cognitive and Self-regulatory Mechanisms of Obesity Study (COSMOS): Study protocol for a randomized controlled weight loss trial examining change in biomarkers, cognition, and self-regulation across two behavioral treatments. Contemp Clin Trials. 2018 Mar;66:20-27. doi: 10.1016/j.cct.2017.12.010. Epub 2017 Dec 22. PMID 29274893